CLINICAL TRIAL: NCT00796666
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Efficacy And Safety Study Of Monotherapy Sitaxsentan Sodium Versus Combination Therapy With Sitaxsentan Sodium And Sildenafil Citrate In Subjects With Pulmonary Arterial Hypertension Who Have Completed Study B1321001 (NCT00795639)
Brief Title: Study Looking at Combination Therapy (Sitaxsentan+Sildenafil) Vs. Monotherapy (Sitaxsentan Alone) SR-PAAS -Sitaxsentan Efficacy And Safety Trial With A Randomized Prospective Assessment Of Adding Sildenafil
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Safety Issue: The trial was prematurely terminated on Dec 9, 2010, due to safety concerns, specifically new emerging evidence of hepatic injury.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1321003
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Hypertension
Keywords: endothelin receptor antagonist (ETRA); Sitaxsentan
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — sitaxsentan; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitaxsentan and Placebo (Experimental): Monotherapy arm
  Interventions: Drug: Sitaxsentan
- Sitaxsentan and Sildenafil (Experimental): Combination treatment
  Interventions: Drug: Sitaxsentan and Sildenafil

INTERVENTIONS:
Drug: Sitaxsentan — Sitaxsentan = 100 mg tablet administered orally, once daily Sildenafil placebo = 1 tablet administered orally, three times a day
  Arms: Sitaxsentan and Placebo
Drug: Sitaxsentan and Sildenafil — Sitaxsentan = 100 mg tablet administered orally, once daily plus Sildenafil = 20 mg tablet administered orally, three times a day
  Arms: Sitaxsentan and Sildenafil

SUMMARY:
As monotherapy for pulmonary arterial hypertension (PAH) begins to fail additional therapies are introduced. Although co-administration of sitaxsentan and sildenafil is well tolerated the controlled safety/efficacy database of the combination is limited.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in B1321001 (NCT00795639) and completed the 12-week study as planned.

Exclusion Criteria:

* Treated with an investigational drug, other than sitaxsentan sodium in B1321001 (NCT00795639), or device that has not received regulatory approval within the 30 days prior to Baseline/Day 1 or during the study.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2009-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (12):
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Weston, Florida
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Pfizer Investigational Site, Buenos Aires, Argentina
- Pfizer Investigational Site, Sofia, Bulgaria
- Pfizer Investigational Site, Temuco, Chile
- China (3):
  - Pfizer Investigational Site, Changsha, Hunan
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai
- Pfizer Investigational Site, Bogotá, Cundinamarca, Colombia
- Pfizer Investigational Site, Prague, Czechia
- India (7):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Surat, Gujarat
  - Pfizer Investigational Site, Vadodara, Gujarat
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Coimbatore, Tamil Nadu
  - Pfizer Investigational Site, Madurai, Tamil Nadu
- Pfizer Investigational Site, George Town, Pulau Pinang, Malaysia
- Pfizer Investigational Site, Monterrey, Nuevo León, Mexico
- Pfizer Investigational Site, Lima, Peru
- Romania (2):
  - Pfizer Investigational Site, Cluj-Napoca, Romania
  - Pfizer Investigational Site, Iași
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Pfizer Investigational Site, Belgrade, Serbia
- Pfizer Investigational Site, Johannesburg, South Africa
- Pfizer Investigational Site, Bangkoknoi, Bangkok, Thailand
- Pfizer Investigational Site, Istanbul, Fatih, Turkey (Türkiye)
- Pfizer Investigational Site, Kyiv, Ukraine

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321003&StudyName=Study%20Looking%20at%20Combination%20Therapy%20%28Sitaxsentan+Sildenafil%29%20Vs.%20Monotherapy%20%28Sitaxsentan%20Alone%29%20SR-PAAS%20-Sitaxsentan%20Efficacy%20And%20Safety

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who successfully completed treatment in study B1321001 (NCT00795639).
Groups:
- Sitaxsentan and Placebo: Sitaxsentan sodium (100 milligrams [mg]) orally once daily and placebo orally three times a day (TID)
- Sitaxsentan and Sildenafil: Sitaxsentan sodium (100 mg) orally once daily and sildenafil citrate (20 mg) TID
Period: Overall Study
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Started | 67 | 64
Treated | 66 | 64
Randomized and Not Treated | 1 | 0
Completed | 0 | 0
Not Completed | 67 | 64
Not completed — Death | 2 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 7 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 1 | 0
Not completed — Terminated by sponsor | 53 | 55
Not completed — Randomized and not treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Customized [Number; unit: participants]
  less than 18 years | 1 | 0 | 1
  18-44 years | 38 | 41 | 79
  45-64 years | 20 | 18 | 38
  >= 65 years | 8 | 5 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 49 | 104
  Male | 12 | 15 | 27
World Health Organization (WHO) Functional Classification [Number; unit: number] — WHO Pulmonary Atrial Hypertension (PAH) Functional Classification: I (no limitation on physical activity), II (slight limitation on ordinary physical activity), III (marked limitations on physical activity comfortable at rest) and IV (unable to carry out any physical activity without symptoms, dyspnea and fatigue present at rest).
  number
    Functional Class I | 0 | 0 | 0
    Functional Class II | 12 | 11 | 23
    Functional Class III | 55 | 52 | 107
    Functional Class IV | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinical Worsening (TTCW)
Description: Clinical worsening defined as time between first dose of study drug and occurrence of death; or heart-lung/lung transplant; or hospitalization for worsening pulmonary atrial hypertension (PAH); or atrial septostomy; or withdrawal due to addition of chronic medications for treatment of worsening PAH: prostacyclin/prostacyclin analogues/phosphodiesterase-5inhibitors/alternative endothelin receptor antagonists/intravenous inotropes; or increase of calcium channel blockers or oxygen. TTCW measured as duration between study's first dose date in and date when first clinical worsening event occurs.
Time Frame: Baseline, Weeks 12, 24 or Early Termination (ET)
Population: Intent-to-Treat population (ITT): all participants who were randomized
Measure: Median (Full Range); unit: Days
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 67 | 64
Days | NA [123 to 356] — Not applicable (NA). Median TTCW not calculated unless at least 50 percent of participants in each treatment group had a clinical worsening event. | NA [119 to 409] — Not applicable (NA). Median TTCW not calculated unless at least 50 percent of participants in each treatment group had a clinical worsening event.
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Test type: Superiority or Other; p = 0.5416, Log Rank; Cox Proportional Hazard = 0.8616, 95% CI 2-sided [0.602 to 1.233]

2. Secondary Outcome: Change From Baseline in the Total Distance Walked During 6 Minute Walk Distance (6MWD)
Description: 6 MWD was the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed. Continuous pulse oximetry was conducted during the test for safety. Change from baseline = score at Week x - score at baseline.
Time Frame: Baseline to Weeks 12 and 24
Population: ITT; N=number of participants analyzed; Missing values at Weeks 12 and 24 imputed with the last non-missing 6MWD based on the last observation carried forward (LOCF) method
Measure: Mean (Standard Deviation); unit: meters (m)
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 66 | 64
meters (m)
  Baseline | 350.9 (74.47) | 354.7 (79.88)
  Change at Week 12 | -6.9 (71.00) | 23.2 (56.49)
  Change at Week 24 | -5.4 (62.74) | 17.5 (66.84)
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.0049, ANCOVA — P-value was based on the analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO Functional Class (FC) as fixed effects and baseline 6 Minute Walk Distance (6MWD) as a covariate

3. Secondary Outcome: Change From Baseline in World Health Organization (WHO) Functional Class in Participants With PAH at Weeks 12, 24, 48
Description: WHO PAH Functional Classification of physical activity limitations: I (no limitation), II (slight limitation), III (marked limitations, comfortable at rest) and IV (unable to carry out any physical activity without symptoms). The change from baseline in WHO class was classified as Improved (decrease in functional class), No Change (functional class stayed the same), and Worsened (functional class increased). The change from baseline in WHO functional class at Week X was summarized with frequency count and percentage in each category based on imputed data for missing values at Week X.
Time Frame: Baseline, Weeks 12, 24 or ET
Population: ITT
Measure: Number; unit: participant
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 67 | 64
participant
  Week 12 Improvement | 14 | 14
  Week 12 No Change | 52 | 49
  Week 12 Deterioration | 1 | 1
  Week 24 Improvement | 13 | 16
  Week 24 No Change | 53 | 47
  Week 24 Deterioration | 1 | 1
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.8223, Cochran-Mantel-Haenszel — Missing values at Week 12 and Week 24 were imputed with the last non-missing WHO FC based on the last observation carried forward (LOCF) method; Cochran-Mantel-Haenszel (CMH) test used modified ridit scores and the p-value corresponding to the ANCOVA (row mean scores) statistic was reported

4. Secondary Outcome: Change in 36-Item Short-Form Health Survey (SF-36) From Baseline at Weeks 12, 24 and 48 - Physical Functioning Domain
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Change from baseline = Physical Functioning score at Week x minus score at baseline.
Time Frame: Baseline, Weeks 12, 24 and ET
Population: ITT; N=number of participants analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 66 | 63
units on a scale
  Baseline | 37.7 (8.95) | 37.0 (9.95)
  Change at Week 12 | -0.3 (6.97) | 2.9 (6.26)
  Change at Week 24 | 0.7 (6.78) | 3.7 (8.16)
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-3.13 to 1.20], Standard Error of Mean 1.09 — Least squared (LS) mean and p-value based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Physical Functioning Score as a covariate
Statistical Analysis 2: Comparison: Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 2.33, 95% CI 2-sided [0.31 to 4.36], Standard Error of Mean 1.02 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.0094, ANCOVA — P-value based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Physical Functioning Score as a covariate

5. Secondary Outcome: Change in 36-Item Short-Form Health Survey (SF-36) From Baseline at Weeks 12, 24 and 48 - Role Limitations Due to Physical Health Problems Domain
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Change from baseline = Role Limitations Due to Physical Health Problems score at Week x minus score at baseline.
Time Frame: Baseline, Weeks 12, 24 or ET
Population: ITT; N=number of participants analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 66 | 62
units on a scale
  Baseline | 37.9 (10.21) | 36.8 (9.85)
  Change at Week 12 | -2.2 (9.72) | 1.5 (7.08)
  Change at Week 24 | 0.7 (7.63) | 2.6 (7.87)
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-3.92 to 1.20], Standard Error of Mean 1.29 — LS mean based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Role Limitations Due to Physical Health Problems Score as a covariate
Statistical Analysis 2: Comparison: Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 1.99, 95% CI 2-sided [-0.38 to 4.35], Standard Error of Mean 1.19 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.0244, ANCOVA — P-value based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Role Limitations Due to Physical Health Problems Score as a covariate

6. Secondary Outcome: Change in 36-Item Short-Form Health Survey (SF-36) From Baseline at Weeks 12, 24 and 48 - Bodily Pain Domain
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Change from baseline = Bodily Pain score at Week x minus score at baseline.
Time Frame: Baseline, Weeks 12, 24 or ET
Population: ITT; N=number of participants analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 66 | 62
units on a scale
  Baseline | 46.9 (10.19) | 45.1 (10.37)
  Change at Week 12 | -0.7 (7.96) | 3.1 (9.91)
  Change at Week 24 | -1.6 (8.04) | 0.8 (9.86)
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-3.78 to 2.04], Standard Error of Mean 1.46 — LS mean based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Bodily Pain Score as a covariate
Statistical Analysis 2: Comparison: Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 2.24, 95% CI 2-sided [-0.41 to 4.90], Standard Error of Mean 1.34 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.0624, ANCOVA — P-value based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Bodily Pain Score as a covariate

7. Secondary Outcome: Change in 36-Item Short-Form Health Survey (SF-36) From Baseline at Weeks 12, 24 and 48 - General Health Domain
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Change from baseline = General Health score at Week x minus score at baseline.
Time Frame: Baseline, Weeks 12, 24 or ET
Population: ITT; N=number of participants analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 66 | 63
units on a scale
  Baseline | 38.8 (9.69) | 38.9 (9.35)
  Change at Week 12 | -0.5 (6.73) | 2.1 (7.86)
  Change at Week 24 | 0.5 (7.68) | 2.8 (9.10)
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-2.57 to 2.06], Standard Error of Mean 1.17 — LS mean based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FCvas fixed effects and baseline General Health Score as a covariate
Statistical Analysis 2: Comparison: Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 2.65, 95% CI 2-sided [0.48 to 4.82], Standard Error of Mean 1.09 — LS mean based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline General Health Score as a covariate
Statistical Analysis 3: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.0324, ANCOVA — P-value based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline General Health Score as a covariate

8. Secondary Outcome: Change in 36-Item Short-Form Health Survey (SF-36) From Baseline at Weeks 12, 24 and 48 - Vitality Domain
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Change from baseline = Vitality score at Week x minus score at baseline.
Time Frame: Baseline, Weeks 12, 24 or ET
Population: ITT; N=number of participants analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 66 | 62
units on a scale
  Baseline | 46.6 (9.23) | 45.7 (10.47)
  Change at Week 12 | -0.7 (8.22) | 3.2 (8.74)
  Change at Week 24 | 1.4 (7.84) | 2.9 (9.80)
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-2.10 to 2.97], Standard Error of Mean 1.28 — LS mean based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Vitality Score as a covariate
Statistical Analysis 2: Comparison: Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 4.09, 95% CI 2-sided [1.74 to 6.45], Standard Error of Mean 1.19 — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.0136, ANCOVA — P-value based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Vitality Score as a covariate

9. Secondary Outcome: Change in 36-Item Short-Form Health Survey (SF-36) From Baseline at Weeks 12, 24 and 48 - Social Functioning Domain
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Change from baseline = Social Functioning score at Week x minus score at baseline.
Time Frame: Baseline, Weeks 12, 24 or ET
Population: ITT; N=number of participants analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 66 | 62
units on a scale
  Baseline | 41.8 (11.15) | 41.5 (10.19)
  Change at Week 12 | 0.4 (9.72) | 2.5 (8.48)
  Change at Week 24 | 0.9 (10.56) | 0.7 (9.61)
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-2.33 to 3.23], Standard Error of Mean 1.40 — LS mean based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Social Functioning Score as a covariate
Statistical Analysis 2: Comparison: Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 2.73, 95% CI 2-sided [0.14 to 5.32], Standard Error of Mean 1.31 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.1582, ANCOVA — P-value based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Social Functioning Score as a covariate

10. Secondary Outcome: Change in 36-Item Short-Form Health Survey (SF-36) From Baseline at Weeks 12, 24 and 48 - Role Limitation Due to Emotional Problems Domain
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Change from baseline = Role Limitations Due to Emotional Problems score at Week x minus score at baseline.
Time Frame: Baseline, Weeks 12, 24 or ET
Population: ITT; N=number of participants analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 66 | 62
units on a scale
  Baseline | 40.1 (12.30) | 37.7 (11.28)
  Change at Week 12 | -1.9 (10.91) | 0.9 (8.84)
  Change at Week 24 | -0.5 (9.72) | -1.2 (10.09)
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-3.09 to 3.18], Standard Error of Mean 1.58 — LS mean based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Role Limitation Due to Emotional Problems Score as a covariate
Statistical Analysis 2: Comparison: Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 2.27, 95% CI 2-sided [-0.62 to 5.16], Standard Error of Mean 1.46 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.2161, ANCOVA — P-value based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Role Limitation Due to Emotional Problems Score as a covariate

11. Secondary Outcome: Change in 36-Item Short-Form Health Survey (SF-36) From Baseline at Weeks 12, 24 and 48 - Mental Health Domain
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Change from baseline = Mental Health score at Week x minus score at baseline.
Time Frame: Baseline, Weeks 12, 24 or ET
Population: ITT; N=number of participants analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 66 | 62
units on a scale
  Baseline | 45.0 (11.60) | 44.5 (11.50)
  Change at Week 12 | 0.2 (9.65) | 2.5 (10.92)
  Change at Week 24 | 1.6 (9.26) | 1.3 (11.60)
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [-1.61 to 4.50], Standard Error of Mean 1.54 — LS mean based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Mental Health Score as a covariate
Statistical Analysis 2: Comparison: Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 3.66, 95% CI 2-sided [0.82 to 6.50], Standard Error of Mean 1.43 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.2087, ANCOVA — P-value based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Mental Health Score as a covariate

12. Secondary Outcome: Change in 36-Item Short-Form Health Survey (SF-36) From Baseline at Weeks 12, 24 and 48 - Composite Mental Health
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Change from baseline = Composite Mental Health score at Week x minus score at baseline.
Time Frame: Baseline, Weeks 12, 24 or ET
Population: ITT; N=number of participants analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 66 | 62
units on a scale
  Baseline | 45.1 (11.98) | 43.9 (11.29)
  Change at Week 12 | -0.4 (8.67) | 1.6 (9.36)
  Change at Week 24 | 0.3 (8.45) | -0.6 (10.16)
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 1.18, 95% CI 2-sided [-1.21 to 3.58], Standard Error of Mean 1.21 — LS mean based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Composite Mental Health Score as a covariate
Statistical Analysis 2: Comparison: Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 2.71, 95% CI 2-sided [0.37 to 5.05], Standard Error of Mean 1.18 — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.2897, ANCOVA — P-value based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Composite Mental Health Score as a covariate

13. Secondary Outcome: Change in 36-Item Short-Form Health Survey (SF-36) From Baseline at Weeks 12, 24 and 48 - Composite Physical Health
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Change from baseline = Composite Physical Health score at Week x minus score at baseline.
Time Frame: Baseline, Weeks 12, 24 or ET
Population: ITT; N=number of participants analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 66 | 62
units on a scale
  Baseline | 39.7 (8.01) | 39.1 (7.97)
  Change at Week 12 | -0.1 (6.79) | 2.4 (5.54)
  Change at Week 24 | -0.1 (6.49) | 3.1 (6.34)
Statistical Analysis 1: Comparison: Sitaxsentan and Placebo; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-2.05 to 1.38], Standard Error of Mean 0.86 — LS mean based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Composite Physical Health Score as a covariate
Statistical Analysis 2: Comparison: Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 2.14, 95% CI 2-sided [0.46 to 3.82], Standard Error of Mean 0.85 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Sitaxsentan and Placebo vs Sitaxsentan and Sildenafil; Baseline to Week 12; Test type: Superiority or Other; p = 0.0179, ANCOVA — P-value based on analysis of covariance on change from baseline with B1321003 treatment, B1321001 (NCT00795639) treatment, B1321003 Baseline WHO FC as fixed effects and baseline Composite Physical Health Score as a covariate

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sitaxsentan and Placebo | Sitaxsentan and Sildenafil
Serious Adverse Events (participants affected / at risk) | 14/66 | 15/64
Other Adverse Events (participants affected / at risk) | 26/66 | 28/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan and Placebo (N=66) | Sitaxsentan and Sildenafil (N=64)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac asthma (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 3 | 1
Torsade de pointes (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Malaria (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 3 | 3
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan and Placebo (N=66) | Sitaxsentan and Sildenafil (N=64)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 2 | 2
Fatigue (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 6 | 5
Pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 3 | 2
Bronchitis (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 2
Blood creatinine increased (Investigations) | 2 | 0
Blood pressure decreased (Investigations) | 0 | 2
Venous pressure jugular increased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Dizziness (Nervous system disorders) | 6 | 1
Headache (Nervous system disorders) | 2 | 7
Syncope (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Hypotension (Vascular disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
Study terminated early by sponsor, no Week 48 information collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.